CLINICAL TRIAL: NCT01058382
Title: Progesterone Support for Frozen Embryo Transfer: Intramuscular Versus Vaginal Suppository - A Prospective, Randomized, Controlled Trial
Brief Title: Progesterone Support of FET
Acronym: FETProg
Status: Completed | Type: Observational
Sponsor: Charles Coddington (Other)
Responsible Party: Sponsor-Investigator, Charles Coddington, Charles C. Coddington MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Other Study IDs: 09-008006
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Frozen Embryo Pregnancy Rate
Keywords: FET; Progesterone Support; Frozen Embryo Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Progesterone Vaginal Suppositories
  Interventions: Drug: Progesterone Vaginal Suppositories
- Intramuscular Progesterone-in-Oil
  Interventions: Drug: Intramuscular Progesterone-in-Oil

INTERVENTIONS:
Drug: Progesterone Vaginal Suppositories — Progesterone Vaginal Suppositories 200 mg three times daily for 10 weeks following embryo transfer
  Groups: Progesterone Vaginal Suppositories
Drug: Intramuscular Progesterone-in-Oil — Progesterone-in-Oil 50 mg IM once daily for 10 weeks following embryo transfer
  Groups: Intramuscular Progesterone-in-Oil

SUMMARY:
There have been two very common forms of progesterone administration that have been used during ovulation induction, in vitro fertilization (IVF) and embryo transfers. There are currently no randomized clinical trials to demonstrate which method of progesterone administration is more effective for frozen embryo transfer. We raise the question: Is there a difference between the two accepted methods of progesterone administration, intramuscular and vaginal suppositories, for frozen embryo transfer? Studies for fresh embryo transfer after in vitro fertilization, have demonstrated that there is not a difference between the two methods of progesterone administration. We will evaluate the question for frozen embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Females < 50 years of age
* Having frozen embryo transfer at Mayo Clinic
* Embryos have been created prior to age 42
* Willing to be randomized to either method of progesterone administration

Exclusion Criteria:

* Diagnosis of severe medical illness
* Uterine lesions affecting the cavity or endometrium
* Uterine anomaly
* Presence of hydrosalpinx
* Extreme difficulty with embryo transfer

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women having a frozen embryo transfer.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | 3 years

SECONDARY OUTCOMES:
Implantation rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Coddington, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States